CLINICAL TRIAL: NCT03580421
Title: Cost-utility, Safety and Feasibility of Ambulatory Surgery Versus Traditional Pathway in the Management of Endometrial Cancer: a Multicentre, Prospective and Randomised Study
Brief Title: Cost-utility of Ambulatory Surgery in the Management of Endometrial Cancer(AMBU-ENDO)
Acronym: AMBU-ENDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ecole d'econmie de Paris (PSE)-Hospinnomics (Unknown); Université Montpellier (Other); Université de Rennes 1 CREM CNRS UMR 6211 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P150966; 2017-A02835-48 (Registry Identifier: ID RCB)
Record Dates: First submitted 2018-06-06; First posted 2018-07-09 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Endometrial Cancer Stage I; Endometrial Cancer Stage II
Keywords: Endometrial Cancer; Health-economics analysis; Ambulatory surgery; QALY; discrete choice experiment
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Ambulatory Surgical Procedures

STUDY DESIGN:
Intervention Model Description: a multicentre, prospective and randomised study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard pathway group (Active Comparator): this group will benefit from standard care including: one surgical consultation, one anesthesia consultation, surgery followed by 2-4 days of hospitalization and most of the time 3 post-operative consultations (M1, M6, M12) during the first operative year
  Interventions: Procedure: standard surgery
- ambulatory pathway group (Experimental): Preoperative and postoperative protocols will be applied for optimizing same-day discharge. Gynaecologists, anaesthetists, and nursing staff will work as a team. A specific anesthesia consultation will focus on ambulatory surgery management. A geriatric evaluation will be offered to women over 70 years old with a score ≤14 according to G8 screening tool. A dietetic evaluation will be offered to women with BMI ≥ 35. A nursing consultation will be offered, as patient and their family preparation prior to ambulatory surgery is important.
  Interventions: Procedure: ambulatory surgery

INTERVENTIONS:
Procedure: ambulatory surgery — total hysterectomy and bilateral salpingo-oophorectomy with or without lymphadenectomy
  Arms: ambulatory pathway group
Procedure: standard surgery — total hysterectomy and bilateral salpingo-oophorectomy with or without lymphadenectomy
  Arms: standard pathway group

SUMMARY:
To date, cost-utility, safety, and feasibility of ambulatory surgery versus traditional pathway in the management of endometrial cancer have never been prospectively assessed.

The investigators hypothesize that ambulatory surgery versus standard pathway in the management of endometrial cancer is both safe, feasible and may impact on patient health-related quality of life.

The main objective of the study is to assess the cost-utility of ambulatory surgery versus standard pathway in the management of endometrial cancer.

A total of 252 consecutive, eligible, consenting patients with a low- and intermediate-risk early stage endometrial cancer will be enrolled from various clinical practice sites within France and patient will randomly be assigned to one of the two surgical management pathways: ambulatory pathway versus standard pathway.

DETAILED DESCRIPTION:
In developed countries, endometrial cancer is the fourth most common cancer in women. Women with stage I disease, representing almost 75% of cases, have an overall survival of 95%. According to the European guidelines, the standard surgical approach for stage I endometrial cancer consists of laparoscopic total hysterectomy and bilateral salpingo-oophorectomy with or without lymphadenectomy. For patients undergoing laparoscopic surgery for gynecological malignancies, most studies report average hospital stays of 1 day after surgery. Patients are commonly kept in the hospital following surgery for pain and nausea control, prolonged bladder catheterization, and observation for surgical complications. However, some recent retrospective studies show that same-day discharge for patients undergoing laparoscopic staging for endometrial cancer is feasible and safe, despite associated comorbidities (i.e., obesity, hypertension, diabetes) related to endometrial cancer.

A short hospital stay decreases the risk of exposure to hospital infections, causes less disruption to the patient's personal life, results in potential cost savings for patients and relatives, as well as for hospitals, and there is positive feedback regarding the social environment of patients as they return rapidly to daily activities and work.

To date, safety, feasibility and cost-utility of ambulatory surgery versus traditional pathway in the management of endometrial cancer have never been prospectively assessed.

The investigators hypothesize that ambulatory surgery versus standard pathway in the management of endometrial cancer is both safe, feasible and may impact on patient health-related quality of life.

The main objective of the study is to assess the cost-utility of ambulatory surgery versus standard pathway in the management of endometrial cancer.

A total of 252 consecutive, eligible, consenting patients with a low, intermediate- and high-risk early stage endometrial cancer will be enrolled from various clinical practice sites within France and patient will randomly be assigned to one of the two surgical management pathways: ambulatory pathway versus standard pathway.

Preoperative and postoperative protocols (including geriatric and dietetic evaluation, and anesthesia and nursing consultation) will be applied for optimizing same-day discharge of patients randomly assigned to ambulatory surgery.

Data will be collected in conjunction with usual care visit, 1 month after initial surgery.

The economic evaluation will closely follow the 2011 French National Authority for Health (HAS) economic evaluation guidelines and the evaluation proposal will have three complementary parts with a full cooperation between those involved in the evaluation:

First, the economic evaluation will focus on evaluating the cost-utility profile of ambulatory surgery in endometrial cancer in France. This economic evaluation will include a micro-costing study to estimate by direct observation the cost of resources used during the ambulatory pathway, and the total cost of patients' care in each group. The primary endpoint will be the incremental cost-utility ratio using the 30-day health related quality of life. It will be calculated for both groups using health-related quality of life (HRQoL) scores from the EQ-5D and converted to utility scores using French weights. QALYs will be computed at 30 days (primary analysis) using both mortality and HRQoL scores.

Second, the investigators will perform an analysis of patients' and professionals' preferences about ambulatory care pathways. These preferences will be analyzed in depth, using both surveys and recent tools developed in experimental economics. Health care professionals' views and preferences will be collected, using questionnaires and face-to-face interviews both at the beginning of the study (M0). Patients' preferences will be assessed using a Discrete Choice Experiment (DCE) method, which is increasingly used in health economics.

Third, a thorough analysis of the ethical and inequality aspects tied to the development of ambulatory surgery in endometrial cancer will be developed, following the methodological guidance issued in 2013 by the HAS. Special emphasis will be laid on equity issues in the measurement of patients' benefits, using a capability approach (ICECAP-A questionnaire).

Finally, another secondary objective will be to assess the safety and feasibility of ambulatory surgery versus traditional pathway in the management of endometrial cancer, and to validate biomarkers of high risk of nodal involvement in a translational study (complementary budget will be asked for this part).

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age
* Women affiliated to the social security (including CMU)
* Women understanding the French language
* Women with preoperative endometrial biopsy and preoperative MRI to assess disease stage
* Women with stage I or II endometrial cancer according to the 2009 International Federation of Gynecology and Obstetrics (FIGO) classification
* Women eligible for surgery including laparoscopic or vaginal total hysterectomy and bilateral salpingo-oophorectomy with or without nodal staging (i.e., sentinel lymph node biopsy +/- pelvic lymphadenectomy)
* informed consent signed
* pregnant or breast-feeding patient

Exclusion Criteria:

* Nonclinical stage I uterine malignancy
* Women eligible for surgery including nodal staging with para-aortic lymphadenectomy
* Significantly enlarged uterus that prevent intact vaginal removal or will require a laparotomy which may limit ambulatory management (uterine size larger than 10 weeks of gestation)
* Cardiovascular disease (including participants with pacemakers), pulmonary disease
* Estimated life expectancy less than 12 months
* Medically unfit for surgery
* Patient unfit to complete questionnaire
* A history of conversion to laparotomy for lysis of adhésions or significant lysis of adhesions during a surgery
* Previous lymphadenectomy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
the incremental cost-utility ratio | 1 month
  It will be calculated for both groups using health-related quality of life (HRQoL) scores from the EQ-5D and converted to utility scores using French weights

SECONDARY OUTCOMES:
QALYs | 1 month
  QALYs will be computed using both mortality and HRQoL scores
Incidence of Treatment-Emergent Adverse events | 1 month
  number of severe adverse events
Success rate of ambulatory surgery | 1 month
  Rate of women requiring overnight admission
preferences about ambulatory care pathways | inclusion
  Patients' preferences will be assessed using a Discrete Choice Experiment (DCE) method, which is increasingly used in health economics.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffroy CANLORBE, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Lise ROCHAIX, MD PHD, Study Director — Hospinnomics
Locations (9):
- France (9):
  - Service de Chirurgie Gynécologique Obstétrique Reproduction Humaine, Clermont-Ferrand
  - CHIC - Gynécologie-Obstétrique-Maternité, Créteil
  - Service de chirurgie gynécologique, Centre de lutte contre le cancer, Dijon
  - Service de chirurgie gynécologique, Centre Hospitalier Simone Veil, Eaubonne
  - Service de chirurgie gynécologique, hôpital Pitié-salpêtrière, Paris
  - HEGP - Chirurgie Cancérologique Gynécologique et du Sein, Paris
  - Hôpital Bichat-Claude Bernard Gynécologie obstétrique, Paris
  - Service de chirurgie gynécologique, hôpital Tenon, Paris
  - IGR - Comité d'Oncologie Gynécologique, Villejuif